CLINICAL TRIAL: NCT04441307
Title: Strong Foundations: Intervening to Promote Co-Parenting and Reduce Father Hazardous Drinking in Expectant Parents
Brief Title: Promoting Co-Parenting and Reducing Hazardous Drinking in New Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Rochester Institute of Technology (Other); University at Buffalo (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Rina D. Eiden, Professor of Psychology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00003112; 7R01AA027708-02 (NIH); SITE00000607, (Other: Pennsylvania State University - Univ Park Local IRB Study ID)
Record Dates: First submitted 2020-06-14; First posted 2020-06-22 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Parenting; Parent-Child Relations; Drinking, Alcohol; Adjustment
Keywords: Parenting; Couple Relationship; Alcohol and Health
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: In both arms, couples will experience a parenting program for expecting first time parents. In one arm, parents will receive an adapted Family Foundations program. In the other arm, parents will receive an empirically supported community parenting program.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be asked to participate in a parenting program but will not be informed about which arm of the study they have been assigned. To avoid bias in the evaluation of the interventions, outcome assessors will not be informed about which arm of the study participants have been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Foundations (Active Comparator): A community-based parenting education program with individual family check ins will be implemented to all participants assigned to this arm.
  Interventions: Behavioral: Healthy Foundations
- Family Foundations (Experimental): An adapted Family Foundations parenting program for expecting first time parents with individual family check ins will be implemented to all participants assigned to this arm.
  Interventions: Behavioral: Family Foundations

INTERVENTIONS:
Behavioral: Healthy Foundations — Healthy Foundations combines elements of a community-based parent education program with additional information about infant and child development, good parenting practices, parent health behavior, and couple support.
  Arms: Healthy Foundations
Behavioral: Family Foundations — A modified version of Family Foundations, an evidence-based preventive intervention for couples during the transition to parenthood, will be implemented to address several aspects of parent and family adjustment, including parent health behavior, particularly alcohol use, and couple relationship dynamics, to promote a healthy parenting environment.
  Arms: Family Foundations

SUMMARY:
This study aims to understand if a parenting program that helps couples learn to parent as a team and maintain a healthy lifestyle, such as maintaining safer levels of alcohol use, promotes parent and child health and well-being. Programs will be delivered prenatally and postnatally and will include both group classes and individualized sessions. A comprehensive assessment is administered during pregnancy and then at 6 and 12 months of child age. It is hypothesized that targeting intervention during the naturally motivating transition to parenthood may not only provide opportunities for long lasting behavioral change for parents, but also initiate a cascade of protective processes that ultimately reduce risk for negative emotional and behavioral outcomes for children.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant couples who are cohabitating
* Parents are 18 years of age or older
* Health behavior such as moderate to heavy drinking
* English speaking

Exclusion Criteria:

* Plural pregnancy
* Illicit drug use other than cannabis for either parent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Couple Relationship/Co-parenting | 6 months of child age
  Couple relationship will be evaluated through the Co-parenting Relationship Scale. For overall coparenting quality, average responses range from 0 (not true of us/never) to 6 (very true of us/very often). Lower scores indicate worse outcomes.
Parent Adjustment | 6 months of child age
  Parent adjustment will be assessed with self-report on mental health screenings. The Brief Symptom Inventory is a widely used mental health screening measure. Average responses to the listed symptoms range from 0 (not at all) to 4 (extremely) based on how distressing symptoms have been. Higher scores indicate greater intensity of symptoms.
Parent Alcohol Use | 6 months of child age
  Quantity-frequency of alcohol use (Quantity Frequency Index) and frequency of binge drinking (4 or 5 or more on a single occasion) based on the NIAAA standard drink will be assessed. Higher scores indicate greater quantity and frequency of alcohol use and binge drinking, with moderate drinking being defined as up to 1 standard drink per day for women and up to 2 standard drinks per day for men.

SECONDARY OUTCOMES:
Parent-infant Interactions | 6 and 12 months of child age
  Parent-child relations will be measured through the coding of play interaction sessions. Parental warmth, sensitivity, and harshness will be coded during parent-infant interactions. Parents will be asked to spend some time with their infants as they normally would at 6 months. At 12 months, parents will be asked to spend some time with infants as they normally would for the first 5 minutes, and given a series of problem-solving tasks to do with their infants for the next 5 minutes. Warmth (positive affective involvement), sensitivity (e.g., flexibility and contingent responsiveness), and harshness (e.g., intrusive and negative behaviors such as angry/hostile mood and voice, disapproval, and criticism) will be coded based on the global 5-point rating scales of the Early Relational Assessment (Clark, 1999). Higher scores on the rating scales indicate higher frequency of warmth, sensitivity, and harshness.
Infant Self-Regulation | 6 and 12 months of child age
  The Revised Infant Behavior Questionnaire (IBQ-R, Gartstein & Rothbart, 2003) will be used to obtain parent reports of infant reactivity/regulation at 6 and 12 months of infant ages. The scale measures three broad dimensions of behavior Surgency/Extraversion, Negative Affectivity, and Orienting/Regulation. The Surgency/Extraversion dimension includes approach, vocal reactivity, high intensity pleasure, smiling and laughter, activity level, and perceptual sensitivity. The Negative Affectivity dimension includes sadness, distress to limitations, fear, and low falling reactivity. The Orienting/Regulation dimension includes low intensity pleasure, cuddliness, duration of orienting, and soothability. Scores range from 1-7 and higher scores on each dimension reflect higher surgency, negative affect, and regulation. Average of maternal and paternal scores on these three broad dimensions will be included as the final outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Rina D Eiden, PhD, Principal Investigator — Penn State; Stephanie Godleski, PhD, Principal Investigator — Rochester Institute of Technology
Locations (2):
- United States (2):
  - University at Buffalo, Buffalo, New York
  - Rochester Institute of Technology, Henrietta, New York

IPD SHARING:
Plan to Share IPD: No